CLINICAL TRIAL: NCT01046877
Title: A Clinical Study of the Acclarent Tympanostomy Tube Delivery System For The Treatment of Patients Requiring Tympanostomy Tube Insertion For Otitis Media
Brief Title: Singapore Tympanostomy Tube Delivery System Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR005004
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tympanostomy Tube placement (Experimental): Tympanostomy Tube Delivery System (TTDS) used for placement of tympanostomy tubes in patients indicated for such treatment for chronic Otitis Media with Effusion (OME) or recurrent Acute Otitis Media(AOM).
  Interventions: Device: Tympanostomy Tube Delivery System

INTERVENTIONS:
Device: Tympanostomy Tube Delivery System — Placement of the Tympanostomy Tube by the Acclarent Tympanostomy Tube Delivery System (TTDS)
  Other Names: Acclarent Tympanostomy Tube Delivery System

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of the Acclarent Tympanostomy Tube Delivery System (TTDS) in the placement of tympanostomy tubes (TTs) in patients indicated for such treatment for chronic otitis media with effusion (OME) or recurrent acute otitis media (AOM).

ELIGIBILITY:
Inclusion Criteria:

1. >= 1 year of age
2. Diagnosed with either Chronic Otitis Media with Effusion or recurrent Acute Otitis Media and scheduled to undergo bilateral or unilateral tympanostomy tube insertion.
3. Either male or female -

Exclusion Criteria:

1. History of sensitivity or reaction to anaesthesia
2. Markedly atrophic, retracted, atelectatic or perforated tympanic membrane.
3. Otitis externa
4. Active acute otitis media
5. Thickened Tympanic Membrane
6. Thick mucoid effusion (also known as "glue ear")
7. Otitis media pathology requiring T-tubes -

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Tan, MD, Principal Investigator — KK Women's and Children's Hospital, Singapore
Locations (1):
- KK Women's and Children's Hospital Singapore, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive eligible patients presenting to the study site and for whom tube insertion was recommended were offered the opportunity by the investigator to participate in the study.
Groups:
- Tympanic Tube Placement: Tympanostomy Tube Delivery System (TTDS) in the placement of tympanostomy tubes in patients indicated for such treatment for chronic Otitis Media with Effusion (OME) or recurrent Acute Otitis Media(AOM).
  Tympanostomy Tube Delivery System: Placement of the Tympanostomy Tube by the Acclarent Tympanostomy Tube Delivery System (TTDS)
Period: Overall Study
Arm/Group | Tympanic Tube Placement
Started | 25
Completed on Schedule | 6 (Final visit = the earlier of 24 months post-procedure or 12 months after extrusion.)
Completed Study Late | 1 (One completed (evidencing extrusions) at 23.5 mos. Missed 9 mo visit. Exam not possible at 12 mo.)
Completed | 7
Not Completed | 18
Not completed — Exited voluntarily before tube extrusion | 7
Not completed — Exited voluntarily after tube extrusion | 11

BASELINE CHARACTERISTICS:
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Region of Enrollment [Number; unit: participants]
  Singapore | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Ears Treated Successfully With the TTDS in the Absence of Acute Intraprocedural Adverse Events.
Description: TTDS success will be confirmed by the successful delivery of a tube to the tympanic membrane.
Time Frame: Procedural
Population: One subject was missing data on intraprocedural adverse events and is excluded from this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of ears
Units Other Than Participants: ears
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 24
Number analyzed (ears) | 37
percentage of ears | 94.6 [81.8 to 99.3]

2. Secondary Outcome: Percentage of Tympanostomy Tubes Extruded at 12 Months Post Procedure
Time Frame: 12 months
Population: Over the course of 12 months, a total of 17 subjects (25 ears) were assessed at varying follow-up time points as having had tubes extruded. Ears analyzed included those for which a tube was observed to extrude at any follow-up visit and ears that completed the 12 month visit.
Measure: Number (95% Confidence Interval); unit: percentage of tubes
Units Other Than Participants: tubes
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 17
Number analyzed (tubes) | 25
percentage of tubes | 100 [86.3 to 100.0]

3. Secondary Outcome: Percentage of Patent Tubes
Description: This measure assesses the patency (openness or lack of obstruction) of unextruded tubes.
Time Frame: 30 days
Population: One subject (one ear) was lost to follow-up immediately following the procedure.
Measure: Number (95% Confidence Interval); unit: percentage of tubes
Units Other Than Participants: tubes
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 24
Number analyzed (tubes) | 37
percentage of tubes | 94.6 [81.8 to 99.3]

4. Secondary Outcome: Percentage of Patent Tubes
Description: This measure assesses the patency (openness or lack of obstruction) of unextruded tubes.
Time Frame: 3 months
Population: Two subjects were lost to follow-up after the 30 day visit and one subject missed the 3 month visit. One subject was lost to follow-up immediately following the procedure. Thus, only 28 ears of 21 participants had unextruded tubes for assessment of tube patency.
Measure: Number (95% Confidence Interval); unit: percentage of tubes
Units Other Than Participants: tubes
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 21
Number analyzed (tubes) | 28
percentage of tubes | 100 [87.7 to 100.0]

5. Secondary Outcome: Percentage of Patent Tubes
Description: This measure assesses the patency (openness or lack of obstruction) of unextruded tubes.
Time Frame: 6 months
Population: Two subjects lost to follow-up after 3 month visit. Two subjects missed 6 month visit. Two subjects lost to follow-up after 30 day visit. One subject lost to follow-up immediately following procedure. Thus, only 13 ears (= 9 participants) of 18 participants returning at 6 months had unextruded tubes for assessment of patency.
Measure: Number (95% Confidence Interval); unit: percentage of tubes
Units Other Than Participants: tubes
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 9
Number analyzed (tubes) | 13
percentage of tubes | 100 [75.3 to 100.0]

6. Secondary Outcome: Percentage of Patent Tubes
Description: This measure assesses the patency (openness or lack of obstruction) of unextruded tubes.
Time Frame: 9 Months
Population: 3 subjects lost to follow-up after 6 mo visit. 1 subject missed 9 mo visit. 2 subjects lost to follow-up after 3 mo visit. 2 subjects lost to follow-up after 30 day visit. 1 subject lost to follow-up following procedure. Thus, only 3 ears (= 3 participants) of 16 participants returning at 9 mos had unextruded tubes for assessment of patency.
Measure: Number (95% Confidence Interval); unit: percentage of tubes
Units Other Than Participants: tubes
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 3
Number analyzed (tubes) | 3
percentage of tubes | 100 [29.2 to 100.0]

7. Secondary Outcome: Percentage of Ears With Adverse Events
Description: This outcome measure evaluates occurrence of new adverse events since prior follow-up visit. (non-cumulative)
Time Frame: 30 days
Population: One subject was lost to follow-up immediately following the procedure.
Measure: Number (95% Confidence Interval); unit: percentage of ears
Units Other Than Participants: ears
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 24
Number analyzed (ears) | 35
percentage of ears | 2.9 [0.1 to 14.9]

8. Secondary Outcome: Percentage of Ears With Adverse Events
Description: This outcome measure evaluates occurrence of new adverse events since prior follow-up visit. (non-cumulative)
Time Frame: 3 months
Population: One subject was lost to follow-up immediately following the procedure. Two additional subjects were lost to follow-up after the 30 day visit and one subject missed the 30 day visit.
Measure: Number (95% Confidence Interval); unit: percentage of ears
Units Other Than Participants: ears
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 21
Number analyzed (ears) | 33
percentage of ears | 3.0 [0.1 to 15.8]

9. Secondary Outcome: Percentage of Ears With Adverse Events
Description: This outcome measure evaluates occurrence of new adverse events since prior follow-up visit. (non-cumulative)
Time Frame: 6 months
Population: One subject was lost to follow-up immediately following the procedure. Two subjects were lost to follow-up after the 30 day visit. Two additional subjects were lost to follow-up after the 3 month visit and two subject missed the 3 month visit.
Measure: Number (95% Confidence Interval); unit: percentage of ears
Units Other Than Participants: ears
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 18
Number analyzed (ears) | 28
percentage of ears | 0.0 [0.0 to 12.3]

10. Secondary Outcome: Percentage of Ears With Adverse Events
Description: This outcome measure evaluates occurrence of new adverse events since prior follow-up visit. (non-cumulative)
Time Frame: 9 months
Population: One subject was lost to follow-up immediately following the procedure. Two subjects were lost to follow-up after the 30 day visit. Two subjects were lost to follow-up after the 3 month visit. Three additional subjects were lost to follow-up following the 6 month visit and one subject missed the 9 month visit.
Measure: Number (95% Confidence Interval); unit: percentage of ears
Units Other Than Participants: ears
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 16
Number analyzed (ears) | 24
percentage of ears | 0.0 [0.0 to 14.2]

11. Secondary Outcome: Percentage of Ears With Adverse Events
Description: This outcome measure evaluates occurrence of new adverse events since prior follow-up visit. (non-cumulative)
Time Frame: 12 months post procedure
Population: One subject was lost to follow-up following the procedure. 2 subjects were lost to follow-up after the 30 day visit. 2 subjects were lost to follow-up after the 3 month visit. 3 subjects were lost to follow-up following the 6 month visit. 4 subjects were lost to follow-up after the 9 month visit and 2 subjects missed the 12 month visit.
Measure: Number (95% Confidence Interval); unit: percentage of ears
Units Other Than Participants: ears
Arm/Group | Tympanic Tube Placement
Number analyzed (Participants) | 11
Number analyzed (ears) | 17
percentage of ears | 0.0 [0.0 to 19.5]

ADVERSE EVENTS:
Time Frame: Final follow-up visit was the earlier of 24 months post-procedure or 12 months after tube extrusion.
Arm/Group | Tympanic Tube Placement
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tympanic Tube Placement (N=25)
occluded tube/blood in ear (Ear and labyrinth disorders) | 1 (1) — Subject presented with blood in ear and a case of influenza
influenza (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The protocol called for outcome measure assessing patency (openness/lack of obstruction) of unextruded tubes at 12 mos post procedure. Since all tubes had already been extruded by 12 mos, no ears with tubes remained for assessment and it was omitted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days